CLINICAL TRIAL: NCT02031705
Title: Effect of Cavotricuspid Isthmus Ablation in Patients Without History of Typical Flutter During Ablation for Paroxysmal Atrial Fibrillation
Brief Title: Effect of Cavotricuspid Isthmus Ablation in Patients Without History of Typical Flutter During Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yong Seog Oh (Other)
Responsible Party: Sponsor-Investigator, Yong Seog Oh, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTI
Record Dates: First submitted 2013-09-09; First posted 2014-01-09 (Estimated); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Fibrillation; Catheter ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- cavotricuspid isthmus ablation (Active Comparator): Isthmus ablation was performed in paroxysmal atrial fibrillation patients.
  Interventions: Procedure: cavotricuspid isthmus ablation
- control group (Placebo Comparator): Control group was performed no additional cavotricuspid isthmus ablation.
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: cavotricuspid isthmus ablation — Isthmus ablation was performed in paroxysmal atrial fibrillation patients.
  Arms: cavotricuspid isthmus ablation
Procedure: control group — Control group was performed no additional cavotricuspid isthmus ablation.
  Arms: control group

SUMMARY:
It has been demonstrated that successful cavotricuspid isthmus ablation may be effective in preventing paroxysmal atrial fibrillation. However, the effectiveness of only isthmus ablation on atrial fibrillation itself is unclear.

DETAILED DESCRIPTION:
Researchers hypothesized that an organized activation pattern around the tricuspid annulus during atrial fibrillation indicated a mother reentrant circuit that could be terminated by a cavocaval isthmus ablation, thus preventing atrial fibrillation. The objectives of the present study were to evaluate the effectiveness of isthmus ablation in preventing atrial fibrillation and to identify predictors of its success.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled ablation for paroxysmal atrial fibrillation

Exclusion Criteria:

* Typical atrial flutter
* History of artificial tricuspid valve surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2012-07; Primary Completion 2019-06 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Freedom of AF and Af | 1 year after catheter ablation
  1 month, 3 months and 12months after ablation follow up visit and Check the recurrence of atrial fibrillation through EKG,Holter, event recording

CONTACTS AND LOCATIONS:
Overall Officials: SungHwan Kim, MD, Study Director — Seoul St. Mary's Hospital
Locations (1):
- Seoul st. mary's hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim SH, Oh YS, Choi Y, Hwang Y, Kim JY, Kim TS, Kim JH, Jang SW, Lee MY, Joung B, Choi KJ. Long-Term Efficacy of Prophylactic Cavotricuspid Isthmus Ablation during Atrial Fibrillation Ablation in Patients Without Typical Atrial Flutter: a Prospective, Multicentre, Randomized Trial. Korean Circ J. 2021 Jan;51(1):58-64. doi: 10.4070/kcj.2020.0174. Epub 2020 Sep 14. PMID 33150753